CLINICAL TRIAL: NCT03742557
Title: Evaluation of Schemes of Administration of Intravenous Ketamine in Treatment-resistant Depression: Clinical-neuroimaging Correlation
Brief Title: Evaluation of Schemes of Administration of Intravenous Ketamine in Depression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Neurology and Neurosurgery, Mexico (Other)
Responsible Party: Principal Investigator, Rodrigo Pérez Esparza, Medical Sciences Investigator, National Institute of Neurology and Neurosurgery, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 74/18
Record Dates: First submitted 2018-11-08; First posted 2018-11-15 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Treatment Resistant Depression
Keywords: Depression; Ketamine; Treatment-Resistant; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: A double-blind randomized clinical trial (initially) will be performed, followed by an open-label trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Active Comparator): Ketamine 50 MG/ML - at a dose of 0.5 mg/kg IV diluted in 100cc of saline solution 0.9% over 40 minutes.
  The intervention will be done twice weekly for 8 weeks.
  Interventions: Drug: Ketamine 50 MG/ML Injectable Solution, 0.5 mg/kg IV
- Placebo (Placebo Comparator): Saline solution 0.9% over 40 minutes. The intervention will be done twice weekly for 2 weeks, and then patients will receive intervention with ketamine as described above in the Active Comparator.
  Interventions: Drug: Ketamine 50 MG/ML Injectable Solution, 0.5 mg/kg IV

INTERVENTIONS:
Drug: Ketamine 50 MG/ML Injectable Solution, 0.5 mg/kg IV — Ketamine 0.5 mg/kg IV
  Other Names: Ketalar; Anesket

SUMMARY:
Mexico, prevalence reported for major depressive disorder (MDD) is of 7.2%. It is currently in the top 5 causes of disability worldwide. One third of patients will not achieve remission after two treatments, being classified as treatment-resistant. In a neurochemical level, evidence shows dysregulation of the excitatory neurotransmitter Glutamate in patients with MDD. Chronic stress has been related to this dysregulation. Ketamine, has shown to regulate glutamatergic neurotransmission, and specially promote the release and production of neurotrophic factors key in the causes of MDD inhibited by glutamate dysregulation), and allow restoration of areas affected.

Clinical studies of ketamine in MDD have shown robust, durable , and rapid effects (during the first 4-24 hours), allowing a great opportunity for patients who do not achieve benefits from antidepressants or patients with suicidal ideation . These results have been reported in metaanalysis.

To our knowledge, there are no studies using Magnetic Resonance Spectroscopy, in areas related to MDD, after a series of ketamine administrations, which we think may show changes after this chronic administration and explain its antidepressant properties.

Goals: Provide clinical evidence of responseas well as a neurological basis or biomarker of response to a series of ketamine infusions.

DETAILED DESCRIPTION:
1. Background 1.1 Major depressive disorder (MDD) MDD is a clinical syndrome characterized by the presence of low modo, anhedonia, appetite and weight changes, sleep disturbances, psychomotor alterations, fatigue, guilt and low self-esteem, ideas related to death or suicide, and concentration difficulties.

MDD represents one of the first causes of disability worldwide. In Mexico, prevalence is estimated in 7.2% of the population. In accordance to the largest clinical trial of MDD, the STAR*D (Sequenced Treatment Alternatives to Relieve Depression), up to one third of the patients will not achieve remission after 4 treatment strategies. These obligates research of new treatments for MDD and treatment-resistant depression TRD.

1.2 Treatment-resistant Depression (TRD) There is a lack of consensus to define TRD, with multiple criteria used by distinct authors. However, the most used definition is the failure to achieve response or remission after two consecutive treatments at an adequate dose and duration, considering the last episode.

1.3 Physiopathology of MDD. Historically, serotonin and noradrenaline disturbances in production, metabolism and reuptake have been implicated in MDD, as well as dopamine. However, this hypothesis seems insufficient in explaining the lack of immediate response, and the lack of response of up to one third of patients.

It is necessary to understand MDD as a multifactorial disorder (biological, psychological, and environmental agents). At a genetic level, some polymorphisms have been related to the appearance of MDD, such as the gen associated with the glucocorticoid receptor NR3C1, the one related to the monoaminooxidase-A, and the one related to the glucogen kinase-synthase 3. Heredability for MDD has been calculated around 37%.

In a molecular basis, there are three principal factors implicated in the genesis of MDD: neurotrophic factors such as brain-derived neurotrophic factor (BDNF), proinflammatory cytokines (interleukin-1 beta, 6, tumoral necrosis factor alpha), and a dysregulation in the hypothalamus-hypophysis-adrenal axis.

Anatomically speaking, the majority of neuroimaging studies converge in the existence of a hyperactive amygdala, ventral striatum and medial prefrontal cortex to negative stimuli. Among regions of major interest are the amygdala, prefrontal cortex, the cingulate gyrus in its subgenual area and anterior or pregenual area (pgACC), ventral striatum, medial thalamus, posterior cingulate gyrus and anterior insulae.

1.5 Glutamate and GABA in MDD y GABA Glutamatergic and GABAergic dysfunction in affective disorders has increased interest in the last years, evidenced by clinical neuroimaging studies that demonstrate disturbances in such systems in patients with MDD, animal models of stress, and the role of glucocorticoids in the glutamatergic regulation secondary to chronic stress, as well as studies about the action of antidepressants in these systems.

1.6 Magnetic Resonance Spectroscopy H1-MRS in MDD H1-MRS studies coincide with the diminution of glutamate, glutamine and Glx (a composite measure of the previous two) in patients with MDD compared to controls in the pgCCA. Such finding has been correlated with the severity of MDD and anomalous connectivity with the anterior insulae.

Disturbed GABA neurotransmission has been also found in the occipital cortex in patients with MDD and TRD, suggesting a possible biomarker for differential diagnosis. Specifically in TRD patients, Glx in pgACC have been found to be altered, however more studies are needed.

1.7 pgACC in MDD pgACC in MDD refers to the rostral portion of the ACC that englobes the anterior portion of the corpus callosum, nominated sometimes as the medial prefrontal cortex. It comprises Brodmann's areas 24, 25, 32 and 33. The pgACC corresponds to the area 33. Through models of meta-analytic connectivity, its role in the production of interception and subjective feelings, coordinating responses appropriate to internal and external events along with the insulae, and its involvement in the representation of interoceptive information have been confirmed. It seems also to represent the area in with the distinction of cognition and affect takes place39. Such function is supported by evidence of structures connected to the pgACC (lateral and ventromedial prefrontal cortices, and limbic regions).

pgACC activity has been shown to be a predictor of response of some depression treatments such as pharmacological treatments and transcranial magnetic stimulation.

Functional MRI (fMRI), has demonstrated an increased connectivty between pgACC and dorsolateral prefrontal cortex, as well as a diminution in the connectivity of the pgACC and caudate. Such findings may be explained by an intense cognitive control over emotional regulation in MDD patients.

There is evidence of abnormal glutamatergic abnormalities in cerebral activity in resting state in MDD patients, finding a correlation between lower glutamate levels in the pgACC and a diminished connectivity of the same area with the anterior insulae compared to controls through H1-MRS and BOLD techniques.

Because of these findings, it is of great interest for the investigators to study this region in relation to ketamine interventions as an antidepressant therapy.

1.9 Ketamine as an antidepressant Ever since the first clinical study reporting the use of ketamine as an antidepressant for TRD patients, showing a rapid (in hours) and robust (in days) response after a unique administration, the literature has grown exponentially. However, mechanisms of action remain inconclusive.

Its antidepressant properties have been vinculated by ketamine's capacity to stimulate the release and expression of BDNF. Contrary to the result of chronic stress, inhibiting these results, ketamine seems to stimulate it. This molecule is involved in the modulation of neuroplasticity, specifically in the prefrontal cortices. Another of the explanations in a molecular level has been its regulation in the glycogen kinase-synthase 3 (GSK3), required for the pruning and synaptic reconsolidation50. Finally, ketamine has been shown to regulate the lateral habenula (implicated in MDD), probably also explaining its role in the down-regulation of monoamines.

Its clinical effects make ketamine a candidate to solve problems related to MDD in public health, confirmed by various systematic reviews and meta-analysis.

There are clinical trials reporting the efficacy of repeated administrations of ketamine (from 7 days up to 83 days after the last administration) with IV ketamine and intranasal esketamine. However, studies vary in the number of interventions, intervals, conditions to continue treatment, times of measurements, follow-up, making it impossible to obtain standardized results. Also, repeated doses have not been reported with H1-MRS technique to explore if there are durable changes after chronic administration of subanesthetic doses of ketamine in MDD.

1.10 Glutamatergic and GABAergic chances in pgACC before ketamine administration H1-MRS data concerning glutamate levels in healthy subjects show that after ketamine administration, there is a significative increase in glutamate in the pgACC, correlating with psychopathology scales such as the PANSS, supporting the idea that ketamine exerts an important effect in the neurotransmission related to its mechanism of action in this region of interest. Such findings propose the difference in this region of interest pre and postinfusion of ketamine and represent an important antecedent for the current proposal. In a similar way, in healthy subjects, hippocampal augments of Glx and a decreased of the fronto-temporal connectivity and temporo-parietal after the administration measured at 10 minutes after ketamine administration has been shown.

When measuring glutamate, Glx and GABA in the pgACC after ketamine in MDD patients, there have been mixed results. Some authors have found a significative increase of the same, correlating with clinical response when measuring during the infusion53. However, using major tesla MRI and measuring the effect of ketamine in glutamate at 24 hours after administration show no differences against placebo. Both findings are discussed concerning the time of measure, concluding that there is a rapid and robust increase, but a transitory one. However these changes do not persist.

To our knowledge no H1-MRS studies after a series of ketamine infusions to know if there are durable changes in glutamate of GABA levels that may explain the durable antidepressant effects of ketamine.

1.11 Experience in the National Institute of Neurology and Neurosurgery (NINN), Mexico Clinical experience with ketamine as an antidepressant and augmentation agent to conventional antidepressants has shown similar clinical results as reported previously, and even have shown longer times until relapse. There is extensive experience in the utilization of H1-MRS in other disorders. The investigators consider that this institution is ideal for the development of the current proposal.

2.1 Key questions

1. Will patients with TRD have a clinical response (50%) after the infusion of ketamine as measured by the Hamilton Depression Rating Scale (HDRS) and the Montgomery-Asberg Depression Rating Scale (MADRS) during the first 24 hours, and different to patients receiving placebo?
2. Will TRD patients presenting response, present a significant increase in Glutamate and GABA in the pgACC measured by H1-MRS 24 hours after the last intervention, compared to the basal measure?
3. Will this response, if achieved, be different than changes in Glutamate and GABA in the pgACC among patients receiving placebo?

3. METHODOLOGY 3.1 Design A double-blind randomized clinical trial will be performed 3.2 Sample During the sample selection, inclusion and exclusion criteria defined afterwards will be used. Sampling will be non-probabilistic in a consecutive case manner. Patients will participate voluntarily after informed consent is achieved.

Subjects treated in the NINN will be divided in two groups:

1. Subjects with TRD, receiving ketamine infusions from start.
2. Subjects with TRD, receiving placebo (saline solution 0.9%), and afterwards

3.3 Procedure

1. Sampling.
2. Previous evaluation:

   1. Psychiatric evaluation (HDRS-17, MADRS).
   2. Medical evaluation
3. Randomization
4. Basal 1H-MRS for GABA:
5. Basal 1H-MRS for Glutamate:

   Similar to the GABA acquisition.
6. Interventions

   1. All interventions will be done as an out-patient basis by a psychiatrist.
   2. A 0.5 mg/kg infusion of ketamine or placebo IV along 40 minutes will be performed. Vigilance will be strict (vital signs, adverse effects, subjective experience, clinimetry).
   3. After every intervention, the patient will be observed for 1 hour or more if considered necessary by the clinician, returning to their normal routine afterward.
   4. Such intervention will be done twice weekly in a prior of 4 weeks (day 1, 4, 8, 11, 15, 19, 23, and 27) for a total of 8 infusions in patients receiving ketamine.

   i. In case of having received placebo, patients will then receive 8 infusions of ketamine.

   ii. In case of having received ketamine, they will continue until completing 8 infusions, and then receive 4 infusions of placebo.
7. Posterior evaluation

   1. Psychiatric evaluation as explained earlier at 4, 24, 72 hours and weekly up to 12 weeks after the last infusion of relapse.
   2. Glutamate and GABA in pgACC measures with the parameters after 10 minutes of starting the infusion, 24 hours after, and 1 week after the last infusion of ketamine or placebo.
8. Follow-up a. 12-week follow-up after last intervention or relapse, after which patients will end participation and their care will continue as usual.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years
2. MDD diagnosis as provided by DSM-5 criteria
3. TRD as defined by failure to achieve response to two consecutive antidepressant therapies at an adequate dose and duration
4. Patients approving inclusion by signing the informed consent

Exclusion Criteria:

1. Comorbidity with other mental and neurological disorders (except generalized anxiety disorder)
2. Substance use disorders at least 3 months prior to enrollment
3. Evidence of structural abnormalities in basal MRI
4. Pregnancy or lactation
5. Hypersensitivity to ketamine
6. Cardiac failure
7. Personal history of psychosis
8. First-degree relatives with history of psychosis
9. Uncontrolled close-angle glaucoma
10. Neurological disease (present)
11. Uncontrolled Hypertension
12. Contraindications for the realization of H1-MRS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Depression Severity Hamilton Depression Rating Scale | 4, 24, 72 hours, weekly up to 12 weeks or until relapse (Change from baseline to each measure)
  Depression Severity (10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe). Higher values represent a worse severity, but not necessarily outcome.
Glutamate | Basal, 10 minutes during intervention, 24 hours after, 4 weeks after (Change from baseline to each measure)
  Glutamate levels in the pgACC basal and after the last intervention with ketamine or placebo
GABA | Basal, 10 minutes during intervention, 24 hours after, 4 weeks after (Change from baseline to each measure)
  GABA levels in the pgACC basal and after the last intervention with ketamine or placebo
Depression Severity Montgomery-Asberg Depression Rating Scale) | 4, 24, 72 hours, weekly up to 12 weeks or until relapse (Change from baseline to each measure). Higher values represent a worse severity, but not necessarily outcome.
  Depression Severity (9-17 = mild, 18-34 = moderate, and ≥ 35 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Pérez-Esparza, M.D., M.Sc., Principal Investigator — National Institute of Neurology and Neurosurgery
Locations (1):
- Instituto Nacional de Neurología y Neurocirugía (National Institute of Neurology and Neurosurgery), Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No
Undecided.

REFERENCES:
- [Background] American Psychiatric Association., American Psychiatric Association. DSM-5 Task Force. Diagnostic and statistical manual of mental disorders : DSM-5. 5th ed. Arlington, VA: American Psychiatric Association; 2013.
- [Background] Moussavi S, Chatterji S, Verdes E, Tandon A, Patel V, Ustun B. Depression, chronic diseases, and decrements in health: results from the World Health Surveys. Lancet. 2007 Sep 8;370(9590):851-8. doi: 10.1016/S0140-6736(07)61415-9. PMID 17826170
- [Background] Conway CR, George MS, Sackeim HA. Toward an Evidence-Based, Operational Definition of Treatment-Resistant Depression: When Enough Is Enough. JAMA Psychiatry. 2017 Jan 1;74(1):9-10. doi: 10.1001/jamapsychiatry.2016.2586. No abstract available. PMID 27784055
- [Background] Berlim MT, Turecki G. What is the meaning of treatment resistant/refractory major depression (TRD)? A systematic review of current randomized trials. Eur Neuropsychopharmacol. 2007 Nov;17(11):696-707. doi: 10.1016/j.euroneuro.2007.03.009. Epub 2007 May 23. PMID 17521891
- [Background] Wijeratne C, Sachdev P. Treatment-resistant depression: critique of current approaches. Aust N Z J Psychiatry. 2008 Sep;42(9):751-62. doi: 10.1080/00048670802277206. PMID 18696279
- [Background] Harmer CJ, Duman RS, Cowen PJ. How do antidepressants work? New perspectives for refining future treatment approaches. Lancet Psychiatry. 2017 May;4(5):409-418. doi: 10.1016/S2215-0366(17)30015-9. Epub 2017 Jan 31. PMID 28153641
- [Background] Boku S, Nakagawa S, Toda H, Hishimoto A. Neural basis of major depressive disorder: Beyond monoamine hypothesis. Psychiatry Clin Neurosci. 2018 Jan;72(1):3-12. doi: 10.1111/pcn.12604. Epub 2017 Oct 19. PMID 28926161
- [Background] Kupfer DJ, Frank E, Phillips ML. Major depressive disorder: new clinical, neurobiological, and treatment perspectives. Lancet. 2012 Mar 17;379(9820):1045-55. doi: 10.1016/S0140-6736(11)60602-8. Epub 2011 Dec 19. PMID 22189047
- [Background] Pérez-Esparza R. Tratamiento farmacológico de la depresión: actualidades y futuras direcciones. Revista de la Facultad de Medicina. 2017;60(5):7-16.
- [Background] Nutt DJ. The neuropharmacology of serotonin and noradrenaline in depression. Int Clin Psychopharmacol. 2002 Jun;17 Suppl 1:S1-12. doi: 10.1097/00004850-200206001-00002. PMID 12369606
- [Result] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Result] Hirschfeld RM. The epidemiology of depression and the evolution of treatment. J Clin Psychiatry. 2012;73 Suppl 1:5-9. doi: 10.4088/JCP.11096su1c.01. PMID 22951236
- [Result] Medina-Mora ME, Borges G, Benjet C, Lara C, Berglund P. Psychiatric disorders in Mexico: lifetime prevalence in a nationally representative sample. Br J Psychiatry. 2007 Jun;190:521-8. doi: 10.1192/bjp.bp.106.025841. PMID 17541113
- [Result] Hock RS, Or F, Kolappa K, Burkey MD, Surkan PJ, Eaton WW. A new resolution for global mental health. Lancet. 2012 Apr 14;379(9824):1367-8. doi: 10.1016/S0140-6736(12)60243-8. No abstract available. PMID 22500865
- [Result] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Result] Kessler RC, Angermeyer M, Anthony JC, DE Graaf R, Demyttenaere K, Gasquet I, DE Girolamo G, Gluzman S, Gureje O, Haro JM, Kawakami N, Karam A, Levinson D, Medina Mora ME, Oakley Browne MA, Posada-Villa J, Stein DJ, Adley Tsang CH, Aguilar-Gaxiola S, Alonso J, Lee S, Heeringa S, Pennell BE, Berglund P, Gruber MJ, Petukhova M, Chatterji S, Ustun TB. Lifetime prevalence and age-of-onset distributions of mental disorders in the World Health Organization's World Mental Health Survey Initiative. World Psychiatry. 2007 Oct;6(3):168-76. PMID 18188442
- [Result] Luppino FS, de Wit LM, Bouvy PF, Stijnen T, Cuijpers P, Penninx BW, Zitman FG. Overweight, obesity, and depression: a systematic review and meta-analysis of longitudinal studies. Arch Gen Psychiatry. 2010 Mar;67(3):220-9. doi: 10.1001/archgenpsychiatry.2010.2. PMID 20194822
- [Result] Espinosa-Aguilar C-A, Zamora-Olvera, Arronte-Rosales, Krug-Llamas, Olivares-Santos, Reyes-Morales, Tapia-Garcia, Garcia-Gonzalez, Doubova. Guía de práctica clínica para el diagnóstico y tratamiento de depresión en los adultos mayores. Salud Mental. 2007;30(6):69-80.
- [Result] Heinze C. Guía clínica para el Manejo de la Depresión. In: Psiquiatría INd, ed. Guías Clínicas para la Atención de Trastornos Mentales. Mexico D.F.2010.
- [Result] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Result] Trivedi MH, Rush AJ, Wisniewski SR, Nierenberg AA, Warden D, Ritz L, Norquist G, Howland RH, Lebowitz B, McGrath PJ, Shores-Wilson K, Biggs MM, Balasubramani GK, Fava M; STAR*D Study Team. Evaluation of outcomes with citalopram for depression using measurement-based care in STAR*D: implications for clinical practice. Am J Psychiatry. 2006 Jan;163(1):28-40. doi: 10.1176/appi.ajp.163.1.28. PMID 16390886
- [Result] Sullivan PF, Daly MJ, O'Donovan M. Genetic architectures of psychiatric disorders: the emerging picture and its implications. Nat Rev Genet. 2012 Jul 10;13(8):537-51. doi: 10.1038/nrg3240. PMID 22777127
- [Result] Duman RS, Aghajanian GK. Synaptic dysfunction in depression: potential therapeutic targets. Science. 2012 Oct 5;338(6103):68-72. doi: 10.1126/science.1222939. PMID 23042884
- [Result] Nugent AC, Diazgranados N, Carlson PJ, Ibrahim L, Luckenbaugh DA, Brutsche N, Herscovitch P, Drevets WC, Zarate CA Jr. Neural correlates of rapid antidepressant response to ketamine in bipolar disorder. Bipolar Disord. 2014 Mar;16(2):119-28. doi: 10.1111/bdi.12118. Epub 2013 Sep 18. PMID 24103187
- [Result] Dantzer R, O'Connor JC, Freund GG, Johnson RW, Kelley KW. From inflammation to sickness and depression: when the immune system subjugates the brain. Nat Rev Neurosci. 2008 Jan;9(1):46-56. doi: 10.1038/nrn2297. PMID 18073775
- [Result] Raison CL, Borisov AS, Majer M, Drake DF, Pagnoni G, Woolwine BJ, Vogt GJ, Massung B, Miller AH. Activation of central nervous system inflammatory pathways by interferon-alpha: relationship to monoamines and depression. Biol Psychiatry. 2009 Feb 15;65(4):296-303. doi: 10.1016/j.biopsych.2008.08.010. Epub 2008 Sep 18. PMID 18801471
- [Result] MacQueen G, Frodl T. The hippocampus in major depression: evidence for the convergence of the bench and bedside in psychiatric research? Mol Psychiatry. 2011 Mar;16(3):252-64. doi: 10.1038/mp.2010.80. Epub 2010 Jul 27. PMID 20661246
- [Result] Greicius MD, Flores BH, Menon V, Glover GH, Solvason HB, Kenna H, Reiss AL, Schatzberg AF. Resting-state functional connectivity in major depression: abnormally increased contributions from subgenual cingulate cortex and thalamus. Biol Psychiatry. 2007 Sep 1;62(5):429-37. doi: 10.1016/j.biopsych.2006.09.020. Epub 2007 Jan 8. PMID 17210143
- [Result] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Result] DiazGranados N, Ibrahim LA, Brutsche NE, Ameli R, Henter ID, Luckenbaugh DA, Machado-Vieira R, Zarate CA Jr. Rapid resolution of suicidal ideation after a single infusion of an N-methyl-D-aspartate antagonist in patients with treatment-resistant major depressive disorder. J Clin Psychiatry. 2010 Dec;71(12):1605-11. doi: 10.4088/JCP.09m05327blu. Epub 2010 Jul 13. PMID 20673547
- [Result] Valentine GW, Mason GF, Gomez R, Fasula M, Watzl J, Pittman B, Krystal JH, Sanacora G. The antidepressant effect of ketamine is not associated with changes in occipital amino acid neurotransmitter content as measured by [(1)H]-MRS. Psychiatry Res. 2011 Feb 28;191(2):122-7. doi: 10.1016/j.pscychresns.2010.10.009. Epub 2011 Jan 12. PMID 21232924
- [Result] Zarate CA Jr, Brutsche NE, Ibrahim L, Franco-Chaves J, Diazgranados N, Cravchik A, Selter J, Marquardt CA, Liberty V, Luckenbaugh DA. Replication of ketamine's antidepressant efficacy in bipolar depression: a randomized controlled add-on trial. Biol Psychiatry. 2012 Jun 1;71(11):939-46. doi: 10.1016/j.biopsych.2011.12.010. Epub 2012 Jan 31. PMID 22297150
- [Result] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Result] Diazgranados N, Ibrahim L, Brutsche NE, Newberg A, Kronstein P, Khalife S, Kammerer WA, Quezado Z, Luckenbaugh DA, Salvadore G, Machado-Vieira R, Manji HK, Zarate CA Jr. A randomized add-on trial of an N-methyl-D-aspartate antagonist in treatment-resistant bipolar depression. Arch Gen Psychiatry. 2010 Aug;67(8):793-802. doi: 10.1001/archgenpsychiatry.2010.90. PMID 20679587
- [Result] Lener MS, Niciu MJ, Ballard ED, Park M, Park LT, Nugent AC, Zarate CA Jr. Glutamate and Gamma-Aminobutyric Acid Systems in the Pathophysiology of Major Depression and Antidepressant Response to Ketamine. Biol Psychiatry. 2017 May 15;81(10):886-897. doi: 10.1016/j.biopsych.2016.05.005. Epub 2016 May 12. PMID 27449797
- [Result] Musazzi L, Treccani G, Mallei A, Popoli M. The action of antidepressants on the glutamate system: regulation of glutamate release and glutamate receptors. Biol Psychiatry. 2013 Jun 15;73(12):1180-8. doi: 10.1016/j.biopsych.2012.11.009. Epub 2012 Dec 28. PMID 23273725
- [Result] Luykx JJ, Laban KG, van den Heuvel MP, Boks MP, Mandl RC, Kahn RS, Bakker SC. Region and state specific glutamate downregulation in major depressive disorder: a meta-analysis of (1)H-MRS findings. Neurosci Biobehav Rev. 2012 Jan;36(1):198-205. doi: 10.1016/j.neubiorev.2011.05.014. Epub 2011 Jun 6. PMID 21672551
- [Result] Price RB, Shungu DC, Mao X, Nestadt P, Kelly C, Collins KA, Murrough JW, Charney DS, Mathew SJ. Amino acid neurotransmitters assessed by proton magnetic resonance spectroscopy: relationship to treatment resistance in major depressive disorder. Biol Psychiatry. 2009 May 1;65(9):792-800. doi: 10.1016/j.biopsych.2008.10.025. Epub 2008 Dec 5. PMID 19058788
- [Result] Hamani C, Mayberg H, Stone S, Laxton A, Haber S, Lozano AM. The subcallosal cingulate gyrus in the context of major depression. Biol Psychiatry. 2011 Feb 15;69(4):301-8. doi: 10.1016/j.biopsych.2010.09.034. Epub 2010 Dec 8. PMID 21145043
- [Result] Drevets WC, Savitz J, Trimble M. The subgenual anterior cingulate cortex in mood disorders. CNS Spectr. 2008 Aug;13(8):663-81. doi: 10.1017/s1092852900013754. PMID 18704022
- [Result] Savitz JB, Rauch SL, Drevets WC. Clinical application of brain imaging for the diagnosis of mood disorders: the current state of play. Mol Psychiatry. 2013 May;18(5):528-39. doi: 10.1038/mp.2013.25. Epub 2013 Apr 2. PMID 23546169
- [Result] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Result] Davey CG, Harrison BJ, Yucel M, Allen NB. Regionally specific alterations in functional connectivity of the anterior cingulate cortex in major depressive disorder. Psychol Med. 2012 Oct;42(10):2071-81. doi: 10.1017/S0033291712000323. PMID 22954259
- [Result] Horn DI, Yu C, Steiner J, Buchmann J, Kaufmann J, Osoba A, Eckert U, Zierhut KC, Schiltz K, He H, Biswal B, Bogerts B, Walter M. Glutamatergic and resting-state functional connectivity correlates of severity in major depression - the role of pregenual anterior cingulate cortex and anterior insula. Front Syst Neurosci. 2010 Jul 15;4:33. doi: 10.3389/fnsys.2010.00033. eCollection 2010. PMID 20700385
- [Result] Mosebach J, Keilhoff G, Gos T, Schiltz K, Schoeneck L, Dobrowolny H, Mawrin C, Muller S, Schroeter ML, Bernstein HG, Bogerts B, Steiner J. Increased nuclear Olig1-expression in the pregenual anterior cingulate white matter of patients with major depression: a regenerative attempt to compensate oligodendrocyte loss? J Psychiatr Res. 2013 Aug;47(8):1069-79. doi: 10.1016/j.jpsychires.2013.03.018. Epub 2013 Apr 21. PMID 23615187
- [Result] Weber M, Motin L, Gaul S, Beker F, Fink RH, Adams DJ. Intravenous anaesthetics inhibit nicotinic acetylcholine receptor-mediated currents and Ca2+ transients in rat intracardiac ganglion neurons. Br J Pharmacol. 2005 Jan;144(1):98-107. doi: 10.1038/sj.bjp.0705942. PMID 15644873
- [Result] Cohen MG, Chan SL, Bhargava HN, Trevor AJ. Inhibition of mammalian brain acetylcholinesterase by ketamine. Biochem Pharmacol. 1974 May 1;23(11):1647-52. doi: 10.1016/0006-2952(74)90377-3. No abstract available. PMID 4847538
- [Result] Smith DJ, Pekoe GM, Martin LL, Coalgate B. The interaction of ketamine with the opiate receptor. Life Sci. 1980 Mar 10;26(10):789-95. doi: 10.1016/0024-3205(80)90285-4. No abstract available. PMID 6246318
- [Result] Smith DJ, Azzaro AJ, Zaldivar SB, Palmer S, Lee HS. Properties of the optical isomers and metabolites of ketamine on the high affinity transport and catabolism of monoamines. Neuropharmacology. 1981 Apr;20(4):391-6. doi: 10.1016/0028-3908(81)90015-0. No abstract available. PMID 7290352
- [Result] Duman RS, Voleti B. Signaling pathways underlying the pathophysiology and treatment of depression: novel mechanisms for rapid-acting agents. Trends Neurosci. 2012 Jan;35(1):47-56. doi: 10.1016/j.tins.2011.11.004. PMID 22217452
- [Result] Yang Y, Cui Y, Sang K, Dong Y, Ni Z, Ma S, Hu H. Ketamine blocks bursting in the lateral habenula to rapidly relieve depression. Nature. 2018 Feb 14;554(7692):317-322. doi: 10.1038/nature25509. PMID 29446381
- [Result] Evans JW, Lally N, An L, Li N, Nugent AC, Banerjee D, Snider SL, Shen J, Roiser JP, Zarate CA Jr. 7T 1H-MRS in major depressive disorder: a Ketamine Treatment Study. Neuropsychopharmacology. 2018 Aug;43(9):1908-1914. doi: 10.1038/s41386-018-0057-1. Epub 2018 Apr 5. PMID 29748628
- [Result] Milak MS, Proper CJ, Mulhern ST, Parter AL, Kegeles LS, Ogden RT, Mao X, Rodriguez CI, Oquendo MA, Suckow RF, Cooper TB, Keilp JG, Shungu DC, Mann JJ. A pilot in vivo proton magnetic resonance spectroscopy study of amino acid neurotransmitter response to ketamine treatment of major depressive disorder. Mol Psychiatry. 2016 Mar;21(3):320-7. doi: 10.1038/mp.2015.83. Epub 2015 Aug 18. PMID 26283639
- [Result] Rowland LM, Bustillo JR, Mullins PG, Jung RE, Lenroot R, Landgraf E, Barrow R, Yeo R, Lauriello J, Brooks WM. Effects of ketamine on anterior cingulate glutamate metabolism in healthy humans: a 4-T proton MRS study. Am J Psychiatry. 2005 Feb;162(2):394-6. doi: 10.1176/appi.ajp.162.2.394. PMID 15677610
- [Result] Fond G, Loundou A, Rabu C, Macgregor A, Lancon C, Brittner M, Micoulaud-Franchi JA, Richieri R, Courtet P, Abbar M, Roger M, Leboyer M, Boyer L. Ketamine administration in depressive disorders: a systematic review and meta-analysis. Psychopharmacology (Berl). 2014 Sep;231(18):3663-76. doi: 10.1007/s00213-014-3664-5. Epub 2014 Jul 20. PMID 25038867
- [Result] Kishimoto T, Chawla JM, Hagi K, Zarate CA, Kane JM, Bauer M, Correll CU. Single-dose infusion ketamine and non-ketamine N-methyl-d-aspartate receptor antagonists for unipolar and bipolar depression: a meta-analysis of efficacy, safety and time trajectories. Psychol Med. 2016 May;46(7):1459-72. doi: 10.1017/S0033291716000064. Epub 2016 Feb 12. PMID 26867988
- [Result] McGirr A, Berlim MT, Bond DJ, Fleck MP, Yatham LN, Lam RW. A systematic review and meta-analysis of randomized, double-blind, placebo-controlled trials of ketamine in the rapid treatment of major depressive episodes. Psychol Med. 2015 Mar;45(4):693-704. doi: 10.1017/S0033291714001603. Epub 2014 Jul 10. PMID 25010396
- [Result] Romeo B, Choucha W, Fossati P, Rotge JY. Meta-analysis of short- and mid-term efficacy of ketamine in unipolar and bipolar depression. Psychiatry Res. 2015 Dec 15;230(2):682-8. doi: 10.1016/j.psychres.2015.10.032. Epub 2015 Oct 30. PMID 26548981
- [Result] Caddy C, Amit BH, McCloud TL, Rendell JM, Furukawa TA, McShane R, Hawton K, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults. Cochrane Database Syst Rev. 2015 Sep 23;(9):CD011612. doi: 10.1002/14651858.CD011612.pub2. PMID 26395901
- [Result] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Result] Vande Voort JL, Morgan RJ, Kung S, Rasmussen KG, Rico J, Palmer BA, Schak KM, Tye SJ, Ritter MJ, Frye MA, Bobo WV. Continuation phase intravenous ketamine in adults with treatment-resistant depression. J Affect Disord. 2016 Dec;206:300-304. doi: 10.1016/j.jad.2016.09.008. Epub 2016 Sep 12. PMID 27656788
- [Result] Singh JB, Fedgchin M, Daly EJ, De Boer P, Cooper K, Lim P, Pinter C, Murrough JW, Sanacora G, Shelton RC, Kurian B, Winokur A, Fava M, Manji H, Drevets WC, Van Nueten L. A Double-Blind, Randomized, Placebo-Controlled, Dose-Frequency Study of Intravenous Ketamine in Patients With Treatment-Resistant Depression. Am J Psychiatry. 2016 Aug 1;173(8):816-26. doi: 10.1176/appi.ajp.2016.16010037. Epub 2016 Apr 8. PMID 27056608
- [Result] Shiroma PR, Johns B, Kuskowski M, Wels J, Thuras P, Albott CS, Lim KO. Augmentation of response and remission to serial intravenous subanesthetic ketamine in treatment resistant depression. J Affect Disord. 2014 Feb;155:123-9. doi: 10.1016/j.jad.2013.10.036. Epub 2013 Oct 29. PMID 24268616
- [Result] Rasmussen KG, Lineberry TW, Galardy CW, Kung S, Lapid MI, Palmer BA, Ritter MJ, Schak KM, Sola CL, Hanson AJ, Frye MA. Serial infusions of low-dose ketamine for major depression. J Psychopharmacol. 2013 May;27(5):444-50. doi: 10.1177/0269881113478283. Epub 2013 Feb 20. PMID 23428794
- [Result] Murrough JW, Perez AM, Pillemer S, Stern J, Parides MK, aan het Rot M, Collins KA, Mathew SJ, Charney DS, Iosifescu DV. Rapid and longer-term antidepressant effects of repeated ketamine infusions in treatment-resistant major depression. Biol Psychiatry. 2013 Aug 15;74(4):250-6. doi: 10.1016/j.biopsych.2012.06.022. Epub 2012 Jul 27. PMID 22840761
- [Result] Daly EJ, Singh JB, Fedgchin M, Cooper K, Lim P, Shelton RC, Thase ME, Winokur A, Van Nueten L, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine Adjunctive to Oral Antidepressant Therapy in Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):139-148. doi: 10.1001/jamapsychiatry.2017.3739. PMID 29282469
- [Result] Stone JM, Dietrich C, Edden R, Mehta MA, De Simoni S, Reed LJ, Krystal JH, Nutt D, Barker GJ. Ketamine effects on brain GABA and glutamate levels with 1H-MRS: relationship to ketamine-induced psychopathology. Mol Psychiatry. 2012 Jul;17(7):664-5. doi: 10.1038/mp.2011.171. Epub 2012 Jan 3. No abstract available. PMID 22212598
- [Result] Kraguljac NV, Frolich MA, Tran S, White DM, Nichols N, Barton-McArdle A, Reid MA, Bolding MS, Lahti AC. Ketamine modulates hippocampal neurochemistry and functional connectivity: a combined magnetic resonance spectroscopy and resting-state fMRI study in healthy volunteers. Mol Psychiatry. 2017 Apr;22(4):562-569. doi: 10.1038/mp.2016.122. Epub 2016 Aug 2. PMID 27480494
- [Result] Perez-Esparza R, Corona T, Ruiz-Garcia RG, Onate-Cadena N, de la Fuente-Sandoval C, Ramirez-Bermudez J. Time until relapse after augmentation with single-dose ketamine in treatment-resistant depression. Psychiatry Clin Neurosci. 2018 Aug;72(8):623. doi: 10.1111/pcn.12675. Epub 2018 Jun 19. No abstract available. PMID 29744959
- [Result] Perez-Esparza R. Ketamine for Treatment-Resistant Depression: a New Advocate. Rev Invest Clin. 2018;70(2):65-7. doi: 10.24875/RIC.18002501. PMID 29718013
- [Result] de la Fuente-Sandoval C, Reyes-Madrigal F, Mao X, Leon-Ortiz P, Rodriguez-Mayoral O, Jung-Cook H, Solis-Vivanco R, Graff-Guerrero A, Shungu DC. Prefrontal and Striatal Gamma-Aminobutyric Acid Levels and the Effect of Antipsychotic Treatment in First-Episode Psychosis Patients. Biol Psychiatry. 2018 Mar 15;83(6):475-483. doi: 10.1016/j.biopsych.2017.09.028. Epub 2017 Oct 10. PMID 29132653
- [Result] de la Fuente-Sandoval C. Potential Regional Differences in GABA Levels in Patients With Psychosis Compared With Control Subjects. Am J Psychiatry. 2016 Jul 1;173(7):734. doi: 10.1176/appi.ajp.2016.16030261. No abstract available. PMID 27363558
- [Result] de la Fuente-Sandoval C, Reyes-Madrigal F, Mao X, Leon-Ortiz P, Rodriguez-Mayoral O, Solis-Vivanco R, Favila R, Graff-Guerrero A, Shungu DC. Cortico-Striatal GABAergic and Glutamatergic Dysregulations in Subjects at Ultra-High Risk for Psychosis Investigated with Proton Magnetic Resonance Spectroscopy. Int J Neuropsychopharmacol. 2015 Sep 12;19(3):pyv105. doi: 10.1093/ijnp/pyv105. PMID 26364273
- [Result] Singh I, Morgan C, Curran V, Nutt D, Schlag A, McShane R. Ketamine treatment for depression: opportunities for clinical innovation and ethical foresight. Lancet Psychiatry. 2017 May;4(5):419-426. doi: 10.1016/S2215-0366(17)30102-5. Epub 2017 Apr 5. PMID 28395988